CLINICAL TRIAL: NCT06379152
Title: Effect of Bilirubin on Prognosis in Heart Failure With Preserved Ejection Fraction
Status: Recruiting | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Other Study IDs: 2024-04-16
Record Dates: First submitted 2024-04-15; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Prognathism
Keywords: Heart Failure with Preserved Ejection Fraction; Bilirubin; Prognosis
MeSH Terms: conditions — Prognathism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DB≤6.8µmol/L: heart failure with preserved ejection fraction patients with direct bilirubn ≤6.8µmol/L
- DB>6.8µmol/L: heart failure with preserved ejection fraction patients with direct bilirubn >6.8µmol/L

SUMMARY:
Factors influencing the prognosis of patients with heart failure with preserved ejection fraction (HFpEF) have been extensively studied. Previous studies have found that elevated serum total bilirubin levels are associated with cardiac death, heart failure readmission, and all-cause mortality in patients with chronic heart failure. However, the relationship between direct bilirubin and prognosis in patients with HFpEF is unclear.

DETAILED DESCRIPTION:
Patients with heart failure with preserved ejection fraction account for approximately 50% of all heart failure patients, have approximately 1.4 hospitalisations per year and an annual mortality rate of approximately 15%. Till now, there have no definitively proven therapies that can reduce their morbidity and mortality, HFpEF Patients have a poor prognosis. The current study found that the prognosis of patients with HFpEF may be related to the heterogeneity of the disease, its various phenotypes and multifactorial pathophysiology, which has not been fully elucidated. The current study found that bilirubin is a risk factor for adverse outcomes of various HFpEF-related complications, but the relationship between direct bilirubin and prognosis of HFpEF has not been reported. Therefore the investigators speculate that direct bilirubin is a predictor of prognosis of HFpEF patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged ≥18 years old；
* Diagnosed with HFpEF.

Diagnostic criteria including:

1. left ventricular ejection fraction ≥ 50%;
2. with the symptoms and/or signs of heart failure;
3. Patients in sinus rhythm：BNP≥35pg/ml and/or NT-proBNP≥125pg/ml；Patients with atrial fibrillation：BNP≥105pg/ml and/or NT-proBNP≥365pg/ml.

Exclusion Criteria:

* LVEF less than 49% at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart failure with preserved ejection fraction (HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The level of direct bilirubin | The day when patients on admission
  The level of direct bilirubin
a composite of heart failure rehospitalization or all-cause mortality | In an average of 3 year after discharge
  a composite of heart failure rehospitalization or all-cause mortality

SECONDARY OUTCOMES:
heart failure rehospitalization | In an average of 3 year after discharge
  heart failure rehospitalization
all-cause mortality | In an average of 3 year after discharge
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No